CLINICAL TRIAL: NCT06930443
Title: Oxygen Consumption, Early Postoperative Hypoperfusion and Organ Injury After Cardio-pulmonary Bypass: a Prospective Observational Study
Brief Title: Oxygen Consumption, Hypoperfusion and Organ Injury After Cardio-pulmonary Bypass
Acronym: VO2-EPOC
Status: Recruiting | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Julia Jakobsson, MD, PhD, Consultant Cardiothoracic anaesthesia and intensive care, Uppsala University Hospital
Other Study IDs: FOU2025-00095; 284709 (Other: Uppsala University Hospital Research Review Board)
Record Dates: First submitted 2025-03-17; First posted 2025-04-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass
Keywords: cardiac surgery; cardiopulmonary bypass; postoperative care
MeSH Terms: interventions — Oxygen Consumption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial and central venous blood gases, blood gases from cardiopulmonary bypass circuit Blood samples for organ injury markers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Oxygen consumption measurement — After arrival to the ICU, prior to cessation of iv anaesthetics and extubation, indirect calorimetry will be performed by connecting a metabolic monitor to the ventilator during a minimum of 20 minutes.

SUMMARY:
The goal of this observational study is to understand how oxygen consumption after heart surgery relates to blood flow problems and organ injury. The study focuses on patients over 18 years old who are having planned heart surgery with a heart-lung machine (cardiopulmonary bypass).

The main questions the study aims to answer are:

1. How does oxygen consumption in the early hours after surgery relate to lactate levels (a sign of low oxygen supply to the tissues)?
2. How is oxygen consumption linked to signs of poor blood flow and organ injury (such as heart, kidney, liver, brain, and gut damage)?

Researchers will measure oxygen consumption after surgery using a technique called indirect calorimetry. They will also track blood flow and oxygen use during surgery and check for signs of organ injury the day after the procedure. The study will include 65 participants. People with certain health conditions, like severe anemia, high lactate levels before surgery, or needing intensive care or extra oxygen supply before surgery, will not be included. By understanding how oxygen consumption relates to blood flow and organ injury, this research may help to better manage patients after heart surgery and reduce complications.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery requiring cardiopulmonary bypass

Exclusion Criteria:

* Combined, redo or annuloplasty procedures
* Surgical procedures involving other vascular cannulation than standard direct, such as bicaval or femoral cannulation
* Preoperative hyperlactatemia (>2mmol/L) or anaemia (Hb <90 g/dL)
* Preoperative need for supplementary oxygen or ICU care
* Consent not obtainable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery at a university hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Difference in oxygen consumption in early postoperative hypoperfusion | 0-4 hours after surgery
  Difference in oxygen consumption (VO2I via indirect calorimetry) in ml min-1 m-2 between patients with and without early hyperlactatemia (>2mmol/L)

SECONDARY OUTCOMES:
Evaluation of hypoperfusion parameters as predictors of postoperative oxygen consumption | 0-24 hours after surgery
  Hypoperfusion parameters will be evaluated as a predictors of postoperative oxygen consumption (VO2I, ml min-1 m-2 via indirect calorimetry).
  Blood gas parameters taken preoperatively and at spaced time-points up to 24 hrs after start of surgery:
  1) Central venous oxygen saturation (ScvO2, %, central venous blood gas), 2) Arterial lactate (mmol/L, arterial blood gas), 3) Base excess (BE, mmol/L, arterial blood gas), 4) Venous-to-arterial CO2 difference (ΔPCO2, mmHg, arterial and central venous blood gas) and its ratio with arterial -central venous oxygen content.
  Clinical variables measured hourly or otherwise specified:
  5) Heart rate (beats/min), 6) Mean arterial pressure (MAP, mmHg), 7) Central venous pressure (CVP, mmHg), 8) Vasopressor or inotrope requirement (Y/N, low-intermediate-high), 9) Urine output (mL/24 hours), and 10) net fluid balance (mL/24 hours).
  Additional explorative data analyses for hypothesis generating purposes can be performed.
Evaluation of oxygen delivery and consumption during cardiopulmonary bypass as predictors of postoperative oxygen consumption | 0-4 hours during and after surgery
  Oxygen delivery (DO2I, ml min-1 m-2) and oxygen consumption (VO2I ml min-1 m-2) will be measured during cardiopulmonary bypass by continuous blood parameter monitoring or calculated by blood oxygen content and pump flow. Both mean levels and repeated measures will be analysed as predictors for postoperative oxygen consumption. Additional explorative data analyses for hypothesis generating purposes can be performed.
Evaluation of organ injury biomarkers as predictors of postoperative oxygen consumption | Preoperative and the day after surgery
  Organ injury markers will be evaluated as predictors for postoperative oxygen consumption. Absolute levels, changes from preoperative values, and above normal predicted value (yes/no) will be used in the analysis.
  Blood sampling preoperatively and the day after surgery.
  1. Renal: Creatinine (mmol L-1), Estimated glomerular filtration rate; eGFR (ml min-1 1.73 m-2):
  2. Cardiac: Troponin T; TnT, creatinine kinase-MB; CK-MB, probrain natriuretic peptide; Nt-proBNP (ng L-1)
  3. Hepatic: Aspartate aminotransferase; ASAT, alanine aminotransferase; ALAT(mikrokat L-1)
  4. Brain: Neurofilament light chain; NFL, Glial fibrillary acidic protein, GFAP (ng L-1)
  5. Gut: Medium chain fatty acids; MCFA, Short chain fatty acids; SCFA, conjugated and non-conjugated bile acids (ng ml-1) Additional explorative data analyses for hypothesis generating purposes can be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Hellgren Johanssson, MD PhD Associate Professor, Study Director — Unit for Cardiothoracic Surgery, Dept. of Surgical Sciences, Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Any data will be carefully reviewed to ensure compliance with GDPR and data sharing regulations before being disclosed.